CLINICAL TRIAL: NCT02505360
Title: Comparaison Biochimique et Histologique Des Cartilages Nasal et Auriculaire Chez le fœtus et le Nouveau-né Porteur de Fente Labiale
Brief Title: Biochemical and Histological Comparison of Nasal and Auricular Cartilage in the Fetus and Newborn With Cleft Lip Carrier
Acronym: CARTOON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-052
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Newborn Cleft Lip and Slot Carrier

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nasal and ear cartilage taken from the newborn (Other): to compare biochemical and histological characteristics of both nasal and ear cartilage taken from the newborn at the time of surgical time cheilorhinoplasty
  Interventions: Other: Measurements of concentration of hyaluronic acid as well as in type 1 collagen and 3

INTERVENTIONS:
Other: Measurements of concentration of hyaluronic acid as well as in type 1 collagen and 3

SUMMARY:
We seek to compare biochemically and histologically the nasal cartilage and ear in the newborn cleft lip and slot carrier in order to improve the quality of care and patient comfort after surgery of cheilorhinoplasty which is the primary treatment slots .

The concentration of hyaluronic acid as well as in type 1 collagen and 3 are assayed by immunohistochemistry and study of mRNA and then they are compared according to the type of cartilage.

This comparison is done on nasal cartilage samples and atrial newborns holders of cleft lip and operated in the neonatal period.

Given the difficulty and constraint of time it takes to reach the 20 subjects of our study , we will also add to our population the stillborn babies before 25SA and newborns who die before the age of 28 days and having had an autopsy.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 0 to 5 weeks with an isolated cleft lip and palate, that is to say non-syndromic, and that will be operated for cheilorhinoplasty neonatal, whose parents have read and understood the document Information and accepted and signed informed consent,
* Children born without life before 25SA and whose parents have read and understood the Information and accepted and signed informed consent for diagnostic purposes permission to autopsy and scientific purposes and / or therapeutic.
* Newborns who died before 28 days of life and whose parents have read and understood the Information and accepted and signed informed consent for diagnostic purposes permission to autopsy and scientific purposes and / or therapeutic.
* Patients And relatives of patients who received clear information and having signed an informed consent,
* Patients Benefiting from a health insurance plan

Exclusion Criteria:

* Patient with no lip slots ( bike palate only or other Tessier slot ) )
* Patient having slots syndromic cleft lip
* Patient whose parents refuse entry into the study.
* Children born without life before 25SA
* Newborns who died after 28 days of life

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Measurements of concentration of hyaluronic acid as well as in type 1 collagen and 3 | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Maxillo-Faciale, Caen, France